CLINICAL TRIAL: NCT04935502
Title: Effects of Home Based Exercises With and Without Posture and Ergonomics Training on Pain and Physical Activity Level Among Students With Musculoskeletal Pain Due to COVID-19 Pandemic: A Randomised Controlled Trial
Brief Title: Home Based Exercises With and Without Posture and Ergonomics Training Among Students During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00254
Record Dates: First submitted 2021-06-14; First posted 2021-06-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal Pain; posture; ergonomic; exercise; Covid-19
MeSH Terms: conditions — Musculoskeletal Pain; Motor Activity; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as accessor of the study would be kept blind of the treatment group to which patient would be allocated.After the complete initial screening process, every recruited patient will be accessed by an independent assessor, expert will use outcome measuring tools. his will be recorded as baseline measurement assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home based exercises with postural and ergonomic training (Experimental): Home based exercises which consist of stretching, strengthening exercises along with postural and ergonomic training will be given to participants for a period of one month by a physiotherapist for 60 minutes via distance education
  Interventions: Other: Home based exercises with postural and ergonomic training
- Home based exercises (Experimental): Home based exercises which consist of stretching and strengthening exercises will be given to participants for a period of one month by a physiotherapist for 60 minutes via distance education.
  Interventions: Other: Home based exercises

INTERVENTIONS:
Other: Home based exercises with postural and ergonomic training — Group A will be treated with stretching and strenghtening exercises for 40 minutes along with postural and ergonomic training for 15 minutes session 3 days/week for 4 week.
  Other Names: Rehabilitation following home based exercises with postural and ergonomic training
  Arms: Home based exercises with postural and ergonomic training
Other: Home based exercises — Group B will be given stretching and strengthening exercises for 40 minutes, every alternate day (3 days per week) for 4 weeks.
  Other Names: Rehabilitation following home based exercises training
  Arms: Home based exercises

SUMMARY:
The aim of this study is to investigate the effect of exercises with and without postural and ergonomic training among the students returning to university after quarantine due to COVID-19.

DETAILED DESCRIPTION:
Postural awareness and ergonomic trainings are approaches that can help to relive pain among patients with Musculoskeletal complaints. The purpose of this study was to investigate the effects of posture and ergonomics training for students receiving distance education during the Covid-19 pandemic on musculoskeletal pain and physical activity level

ELIGIBILITY:
Inclusion Criteria:

1. Participant's using gadget like computer, mobile or laptop for online education during quarantine.
2. Participant's having musculoskeletal pain during COVID-19 quarantine.
3. Prolonged sitting and low physical activity during quarantine.
4. Prolonged exposure of screen more than 6 hours per day due online classes during the quarantine.

Exclusion Criteria:

1. Participant's having musculoskeletal pain before the quarantine.
2. Participant's doing any type of physical activity during quarantine.
3. Participant's taking online classes or any online educational program before quarantine.
4. Participant's with known congenital, inflammatory and infectious conditions of spine.
5. Participant's following any ergonomic recommendations or any postural awareness during and after quarantine.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS). | 4 Weeks
  This pain VAS is unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends and orientated from the left (worst) to the right (best).
Extended Nordic Musculoskeletal (NMQ-E). | 4 Weeks
  This is a subjective instrument that is widely used in clinical settings for patients with musculoskeletal disorders. The Extended Nordic Musculoskeletal Questionnaire is applied to determine the prevalence, severity and impact of musculoskeletal symptoms. The NMQ-E interrogates ache, pain or discomfort experienced in the nine body parts (neck, shoulders, back, elbows, wrists/hands, waist, hips/thighs, knees, ankles/feets)
International Physical Activity Questionnaire Short Form (IPAQ-SF). | 4 weeks
  This is a subjective instrument used for assesses physical activities in the last 7 days by 7 questions. It provides information on the time spent on sitting, walking, moderate activities and intense activities.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No